CLINICAL TRIAL: NCT07156175
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of SAR444336 in Participants With Microscopic Colitis in Clinical Remission With Budesonide
Brief Title: A Study to Investigate the Efficacy and Safety of SAR444336 in Adults With Microscopic Colitis in Clinical Remission
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT18053; 2024-519495-83 (Registry Identifier: CTIS); U1111-1314-5201 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-09-03; First posted 2025-09-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Microscopic Colitis
MeSH Terms: conditions — Colitis, Microscopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SAR444336 (Experimental): Each participant will receive several injections of SAR444336. Budesonide will be taken at the dose administered by the physician.
  Interventions: Drug: SAR444336
- Placebo (Placebo Comparator): Each participant will receive several injections of placebo. Budesonide will be taken at the dose administered by the physician.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR444336 — Pharmaceutical form:Solution for injection -Route of administration:Subcutaneous
  Arms: SAR444336
Drug: Placebo — Pharmaceutical form:Solution for injection -Route of administration:Subcutaneous
  Arms: Placebo

SUMMARY:
This is a parallel, placebo-controlled, multicenter, randomized, double-blind, Phase 2, proof of concept study. The study aims to evaluate the efficacy and safety of SAR444336 in adult participants with microscopic colitis. Participants are required to have a histologically confirmed diagnosis of microscopic colitis, be in clinical remission and be receiving budesonide therapy. The overall study duration is approximately 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed diagnosis of microscopic colitis (including all histological sub-types).
* Receiving budesonide therapy.
* Documented clinical remission from 2 weeks before screening.
* At least 1 microscopic colitis relapse in the last 8 months prior to screening that required treatment with budesonide.
* Body mass index within the range 18 to 35 kg/m2 (inclusive) at screening visit.
* All contraceptive methods used by participants should be consistent with local regulations regarding the methods of contraception.

Exclusion Criteria:

* Significant neutrophilic/eosinophilic infiltration, crypt abscesses, granulomata, or any evidence of IBD other than microscopic colitis.
* Evidence of infectious diarrhea in the 3 months prior to randomization.
* Other active diarrheal conditions or suspicion of drug--induced microscopic colitis at screening, or diarrhea predominant irritable bowel syndrome.
* Any current active viral, bacterial, or fungal infection or any medically relevant infection having occurred within 3 weeks before randomization.
* Previous bowel surgeries.
* Planned surgery while receiving study treatment. Dental surgeries or other types of minor surgery requiring only local anesthetic are allowed.
* Other immunologic disorder, except controlled diabetes or thyroid disorder receiving appropriate treatment.
* Presence or history of drug hypersensitivity associated with eosinophilia in the past 6 months.
* History or presence of alcohol or illicit drug abuse within the past 2 years.
* Excessive consumption of beverages containing xanthine bases.
* History of solid organ transplant.
* Active malignancy, lymphoproliferative disease, or malignancy in remission for less than 2 years, except adequately treated (cured) localized carcinoma in situ of the cervix or ductal breast, or squamous cell carcinoma, or basal cell carcinoma of the skin.
* Have experienced any of the following within 12 months before screening: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association Stage III or IV heart failure.
* Participants with a history or presence of another significant illness such as renal, neurological, ophthalmological, psychiatric, endocrine, cardiovascular, gastrointestinal, hepatic disease, metabolic, pulmonary or lymphatic.
* Live attenuated vaccines within 6 weeks of randomization and during the study.
* Currently receiving or had treatment within 12 months prior to screening with B or T cell depleting agents.
* At screening, have abnormal laboratory values or ECG abnormalities.
* Participants with recent tuberculosis (TB) vaccination or positive TB test results.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-04-08 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with sustained steroid-free clinical remission | up to week 24
  Clinical remission defined as no relapse during the 24-week period.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) | up to week 28
Incidence of study investigational medicinal product (IMP) permanent discontinuations and study withdrawals due to treatment-emergent adverse events (TEAEs) | up to week 28
Plasma concentrations of SAR444336 | through week 24
Incidence of treatment-emergent anti-drug antibody (ADA) against SAR444336 | through week 24

CONTACTS AND LOCATIONS:
Locations (25):
- Belgium (2):
  - Investigational Site Number : 0560002, Ghent
  - Investigational Site Number : 0560001, Leuven
- Denmark (2):
  - Investigational Site Number : 2080003, Aarhus
  - Investigational Site Number : 2080002, Hvidovre
- France (2):
  - Investigational Site Number : 2500001, Créteil
  - Investigational Site Number : 2500003, Pessac
- Germany (5):
  - Investigational Site Number : 2760001, Frankfurt am Main
  - Investigational Site Number : 2760005, Ludwigshafen
  - Investigational Site Number : 2760002, Potsdam
  - Investigational Site Number : 2760003, Tübingen
  - Investigational Site Number : 2760004, Ulm
- Hungary (2):
  - Investigational Site Number : 3480002, Budapest
  - Investigational Site Number : 3480003, Székesfehérvár
- Italy (4):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Investigational Site Number : 380004, Milan, Milano
  - Azienda Ospedale Università Padova, Investigational Site Number : 380001, Padua, Padova
  - Fondazione Policlinico Gemelli IRCCS Roma, Investigational Site Number : 380003, Rome, Roma
  - A.O.U. Città della Salute e della Scienza di Torino, Presidio Molinette, S.C. Gastroenterologia U., Investigational Site Number : 380002, Turin, Torino
- Poland (3):
  - Investigational Site Number : 6160002, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160004, Bydgoszcz
  - Investigational Site Number : 6160003, Warsaw
- Sweden (3):
  - Investigational Site Number : 7520001, Linköping
  - Investigational Site Number : 7520002, Stockholm
  - Investigational Site Number : 7520003, Stockholm
- United Kingdom (2):
  - Investigational Site Number : 8260002, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260001, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT18053 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26835&tenant=MT_SNY_9011